CLINICAL TRIAL: NCT04273633
Title: Ultrasound Supraspinatus Tendon Assessment After 448kilohertz Capacitive Resistive Radiofrequency Stimulation in a Sporty Population.
Brief Title: Ultrasound Supraspinatus Tendon Assessment After 448kilohertz Radiofrequency Stimulation in a Sporty Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, SANTIAGO NAVARRO LEDESMA, UNIVERSITY PROFESSOR, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRMRSPORT
Record Dates: First submitted 2020-02-11; First posted 2020-02-18 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Ultrasonography; Shoulder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus on the dominant shoulder
  Interventions: Device: Monopolar 448 kilohertz radiofrequency stimulation
- Placebo Monopolar Radiofrequency stimulus (Placebo Comparator): To simulate the application of Monopolar Radiofrequency stimulus on the dominant shoulder
  Interventions: Device: Placebo comparator

INTERVENTIONS:
Device: Monopolar 448 kilohertz radiofrequency stimulation — 448kilohertz capacitive resistive monopolar radiofrequency will be applied on the dominant shoulder
  Arms: INTERVENTION
Device: Placebo comparator — To simulate a 448kilohertz capacitive resistive monopolar radiofrequency application on the dominant shoulder
  Arms: Placebo Monopolar Radiofrequency stimulus

SUMMARY:
448kilohertz capacitive resistive monopolar radiofrequency is a novel technique in physiotherapy and its usefulness and clinical relevance is still to be investigated at both clinical practice and also in performance. Current studies show promising results in different musculoskeletal disorders, however there no studies in the assessment of quality soft tissue in sporty population after the used of this technique.

DETAILED DESCRIPTION:
Shoulder pain is is one of the most common musculoskeletal disorders, presenting a high prevalence in primary care centers and sport populations. Many factors have been proposed as the cause of pain, however there are no studies analysing possibilities of preventing shoulder injuries by using a radiofrequency stimulus.

The use of 448kilohertz capacitive resistive monopolar radiofrequency as the focus of the treatment looking for improve the quality of the tissue is still to be explored.

The hypothesis of the present project is that focus treatments on 448kilohertz capacitive resistive monopolar radiofrequency on the shoulder will produce better outcomes in terms of ultrasound assessment measured by quantified elastography, and this will decreased the possibilities of get injured.

The stimulus will be carried out on the shoulder region (suprascapular, axillar, subscapular, long thoracic or pectoralis nerves) and the thoracic region. All interventions will be developed by the same examiner, who is a physiotherapist with 6 years of clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years
* Sporty people with at least 3 days of training per week and presenting an upper limb dominance.

Exclusion Criteria:

* Suffer from any painful shoulder condition.
* History of significant shoulder trauma, such as fracture or ultrasonography
* Clinically suspected partial thickness cuff tear, following the classification of Wiener and Seitz.
* Recent shoulder dislocation in the past two years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in supraspinatus tendon measured by quantified elastography imaging at 3 months | Time Frame: time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)]
  The elastography is obtained when the anatomic image on grayscale ultrasound overlaps parametric color image that expresses the rate of deformity of the tissues, soft tissues tend to develop greater deformity and tissue deformity have lower rigidity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ana González Muñon, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Navarro-Ledesma S, Gonzalez-Munoz A. Short-term effects of 448 kilohertz radiofrequency stimulation on supraspinatus tendon elasticity measured by quantitative ultrasound elastography in professional badminton players: a double-blinded randomized clinical trial. Int J Hyperthermia. 2021;38(1):421-427. doi: 10.1080/02656736.2021.1896790. PMID 33691576